CLINICAL TRIAL: NCT01156636
Title: Pulmonary Hypertension Secondary to Heart Failure With Preserved Systolic Function: a Target of Phosphodiesterase - 5 Inhibition in a 1- Year Duration Study
Brief Title: Phosphodiesterase-5 (PDE5) Inhibition and Pulmonary Hypertension in Diastolic Heart Failure
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: University of Milano, Cardiology (Marco Guazzi PI), University of Milano
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 444-10
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2009-06

CONDITIONS: Pulmonary Hypertension; Diastolic Heart Failure
Keywords: Diastolic Heart Failure; Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure, Diastolic | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil (Active Comparator)
  Interventions: Drug: Sildenafil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — 50 mg 3 times/day for 1 year
  Arms: Sildenafil
Drug: Placebo
  Arms: Placebo

SUMMARY:
Prevalence of heart failure (HF) with left ventricular (LV) diastolic dysfunction and preserved ejection fraction (EF) (HFpEF) is increasing. Prognosis worsens with development of pulmonary vasoconstriction and hypertension (PH) and right ventricular (RV) failure. The investigators aimed at modulating pulmonary vascular tone and RV burden in HFpEF due to high blood pressure (HBP), by using the phosphodiesterase-5 (PDE5) inhibitor sildenafil.

DETAILED DESCRIPTION:
Heart failure (HF) with preserved left ventricular (LV) ejection fraction (EF) (HFpEF) is a public health problem and a major topic in clinical cardiology. Its prevalence, in fact, is increasing and the outcome seems to be similar to that of HF with LV systolic dysfunction (LVSD). Pulmonary hypertension (PH) in HFpEF is highly prevalent and often severe and, like in LVSD (3), is a predictor of morbidity and mortality (4). Because of the thin wall and the distensibility, the right ventricle (RV) is much more vulnerable by an excessive afterload than by preload. The pulmonary circulation is a central determinant of RV afterload, and an increase in impendance to RV ejection, like occurring in LV dysfunction, can easily result in RV failure, tricuspid regurgitation, central venous pressure (CVP) rise. Development of RV failure is unanimously viewed as a predictor of poor prognosis but the underlying mechanisms have not been extensively investigated.

Because of the prevalence and clinical significance of PH secondary to HF, attenuation of the pulmonary vascular tone and of the RV hemodynamic burden has been suggested as a goal to be achieved with HF therapy. Attempts with endothelin receptor antagonists, or prostacyclin analogues, were basically unsuccessful. Experimental models and human studies, showing that in HF nitric oxide (NO) - dependent pulmonary vasodilatation is impaired and pulmonary vascular resistance elevation is at least in part due to pulmonary endothelial dysfunction, have suggested therapeutic strategies with agents that increase NO activity, like nitrates or phosphodiesterase - 5 (PDE5) inhibitors (12-14). The latter agents offer the double advantage of selectively dilating the pulmonary vessels and not producing tachyphylaxis.

In this 1-year duration study, the primary end-point was to probe whether pulmonary hemodynamics and RV performance in HFpEF with PH may be targets of PDE5 inhibition with sildenafil.

ELIGIBILITY:
Inclusion Criteria:

* LVEF >50%
* sinus rhythm and stable clinical condition defined as no changes in therapeutic regimen, or hospitalization in the 6 months preceding recruitment.
* pulmonary artery systolic pressure > 40 mm Hg,

Exclusion Criteria:

* Patients receiving nitrates
* A history of pulmonary disease
* Alternative causes of PH other than cardiac-related
* Renal failure (creatinine > 2mg/dL)
* Anemia
* Pericardial disease
* Cardiac amyloidosis

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-01; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Pulmonary hemodynamics | 1 year

REFERENCES:
- [Derived] Guazzi M, Vicenzi M, Arena R, Guazzi MD. Pulmonary hypertension in heart failure with preserved ejection fraction: a target of phosphodiesterase-5 inhibition in a 1-year study. Circulation. 2011 Jul 12;124(2):164-74. doi: 10.1161/CIRCULATIONAHA.110.983866. Epub 2011 Jun 27. PMID 21709061